CLINICAL TRIAL: NCT04491994
Title: Clearing the Fog: Is HCQ Effective in Reducing COVID-19 progression-a Randomized Controlled Trial
Brief Title: Clearing the Fog: Is Hydroxychloroquine Effective in Reducing COVID-19 Progression
Acronym: COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICEF (Other)
Collaborators: Pak Emirates Military Hospital (Other)
Responsible Party: Principal Investigator, sultan mehmood kamran, Classified Medical specialist, UNICEF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sultan Mehmood Kamran 2
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Results first posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Covid19; Progression
Keywords: COVID-19; viral clearance; , mild infection; disease progression; trial; HCQ
MeSH Terms: conditions — COVID-19; Disease Progression | interventions — Hydroxychloroquine; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomization rules were designed by Dr. Wasim Alamgir together with principal investigators and implemented by an independent statistician who was not involved in data analysis. Stratified random sampling was applied to stratify all eligible patients according to age, gender and comorbidities. Computerized random number generator was used and allocation was done in 2:1 sequence. Cards with each group assignment number randomly generated by computer were placed in sequentially numbered envelopes that were opened as the patients were enrolled
Masking Description: Neither patients, nor investigators, nor statisticians were masked to treatment assignment. Lab staff who performed sampling for PCR, basic blood tests and other routine measurement were unaware of treatment information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (SOC) (No Intervention): Patients selected in supportive arm will be given daily standard doses of oral Vit C (2g), Vit D (alfacalcidiol 1µg), Zinc (50mg) and paracetamol (as required).
- HCQ arm (Experimental): Patients selected in experimental arm will be given Tab HCQ (400mg BD on D0 followed by 200mg BD D1-D5) in addition to supportive treatment
  Interventions: Drug: HCQ

INTERVENTIONS:
Drug: HCQ — Tab HCQ 400mg 12 hourly day 0 followed by tab HCQ 200mg 12 hrly for next 5 days
  Other Names: HCQ + Standard of Care (SOC)
  Arms: HCQ arm

SUMMARY:
Brief Summary: Purpose of this study is to evaluate efficacy of hydroxychloroquine (HCQ) in reducing progression of Corona Virus Disease 2019 (COVID - 19) and achieving viral clearance.

Condition or disease :I COVID-19 ntervention/treatment :Drug: Hydroxychloroquine Sulfate Phase: Phase III

DETAILED DESCRIPTION:
This study explores efficacy of HCQ (400mg BD on D0 and 200mg BD D1-D5) in reducing progression of Mild Covid-19 patients and decreasing viral load.

Participants of study will be randomized 2:1 to receive either Active drug or standard of care (SOC) treatment respectively. We aim to demonstrate reduced COVID-19 progression and early viral clearance in individuals on HCQ therapy.

ELIGIBILITY:
Inclusion Criteria:

* Mild Corona virus disease (COVID-19)
* PCR confirmed infection
* Hospital admitted patients

Exclusion Criteria:

* Moderate, severe and critical COVID-19
* day 0 CRP greater than 6mg/dl, ALC < 1000 or evidence of infiltrates on X-ray chest
* comorbidity with life expectancy less than 6 months
* Contraindications to HCQ therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imran m Fazal, FCPS, Study Director — Pak Emirates Military Hospital (PEMH) Rawalpindi
Locations (1):
- Pak Emirates Military Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
data can be shared on demand in SPSS sheet
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: any time when asked
Access Criteria: by email

REFERENCES:
- [Background] Biot C, Daher W, Chavain N, Fandeur T, Khalife J, Dive D, De Clercq E. Design and synthesis of hydroxyferroquine derivatives with antimalarial and antiviral activities. J Med Chem. 2006 May 4;49(9):2845-9. doi: 10.1021/jm0601856. PMID 16640347
- [Background] Murray JJ, Lee MS. Re: Marmor et al.: American Academy of Ophthalmology Statement: Recommendations on screening for chloroquine and hydroxychloroquine retinopathy (2016 Revision). (Ophthalmology 2016;123:1386-1394). Ophthalmology. 2017 Mar;124(3):e28-e29. doi: 10.1016/j.ophtha.2016.06.062. No abstract available. PMID 28219513
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Zhou D, Dai SM, Tong Q. COVID-19: a recommendation to examine the effect of hydroxychloroquine in preventing infection and progression. J Antimicrob Chemother. 2020 Jul 1;75(7):1667-1670. doi: 10.1093/jac/dkaa114. PMID 32196083
- [Background] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Background] Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends. 2020 Mar 16;14(1):72-73. doi: 10.5582/bst.2020.01047. Epub 2020 Feb 19. PMID 32074550
- [Background] Chen J, Liu D, Liu L, Liu P, Xu Q, Xia L, Ling Y, Huang D, Song S, Zhang D, Qian Z, Li T, Shen Y, Lu H. [A pilot study of hydroxychloroquine in treatment of patients with moderate COVID-19]. Zhejiang Da Xue Xue Bao Yi Xue Ban. 2020 May 25;49(2):215-219. doi: 10.3785/j.issn.1008-9292.2020.03.03. Chinese. PMID 32391667
- [Background] Bhimraj A, Morgan RL, Shumaker AH, Lavergne V, Baden L, Cheng VC, Edwards KM, Gandhi R, Muller WJ, O'Horo JC, Shoham S, Murad MH, Mustafa RA, Sultan S, Falck-Ytter Y. Infectious Diseases Society of America Guidelines on the Treatment and Management of Patients with COVID-19. Clin Infect Dis. 2020 Apr 27:ciaa478. doi: 10.1093/cid/ciaa478. Online ahead of print. PMID 32338708

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment during 10th April to 31st May 2020 at department of Pulmonology, Pakistan Emirates Military Hospital (PEMH) Pakistan.
Pre-assignment Details: 672 confirmed PCR positive cases were assessed for eligibility. 132 did not meet selection criteria and excluded.Later,15 withdrew consent and 5 became symptomatic. During follow up 13 patients were found to be deviated from advised therapy and 7 were lost to follow up yielding a final study population of 500.
Groups:
- Control Group: Standard of care (SOC) treatment comprised of oral Vit C, oral Zinc, oral Vit-D and tablet Paracetamol (for body aches/fever), intravenous fluids, hemodynamic monitoring, and laboratory testing for SARS-CoV-2 and baseline blood parameters.
- Intervention Group: Patients selected in experimental arm will be given standard doses of tab HCQ in addition to standard of care (SOC) treatment. side effects will be monitored
  HCQ: Tab HCQ 400mg 12 hourly day 0 followed by tab HCQ 200mg 12 hrly for next 5 days
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started (15 withdrew consent 5 became symptomatic 13 patients non compliant 7 were lost to follow up) | 180 | 360
Completed | 151 | 349
Not Completed | 29 | 11
Not completed — Withdrawal by Subject | 10 | 5
Not completed — developed fever > 3 days | 4 | 1
Not completed — Protocol Violation | 11 | 2
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Population: sample size calculation was done and 540 patients enrolled
Groups:
- Supportive Arm: Patients selected in supportive arm will be given standard doses of oral Vit C, Vit D, Zinc and panadol
- HCQ Arm: Patients selected in experimental arm will be given standard doses of tab HCQ in addition to supportive treatment. side effects will be monitored
  HCQ: Tab HCQ 400mg 12 hourly day 0 followed by tab HCQ 200mg 12 hrly for next 5 days
- Total: Total of all reporting groups
Arm/Group | Supportive Arm | HCQ Arm | Total
Number analyzed (Participants) | 180 | 360 | 540
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 180 | 360 | 540
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 24 | 34
  Male | 170 | 336 | 506
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Pakistan | 180 | 360 | 540

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression
Description: After start of treatment, development of fever > 101 F for > 72 hours, shortness of breath by minimal exertion (10-Step walk test), derangement of basic lab parameters (ALC < 1000 or raised CRP) or appearance of infiltrates on CXR during course of treatment was labeled as progression irrespective of PCR status
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care (SOC): Standard of care (SOC) treatment comprised of daily oral Vit C (2gms), oral Zinc (50mg), oral Vit-D (alfacalcidol 1ug) and tablet Paracetamol (for body aches/fever), intravenous fluids, hemodynamic monitoring, and laboratory testing for SARS-CoV-2 and baseline blood parameters
- Intervention Group: Patients selected in intervention arm were given HCQ in addition to standard of care treatment. After 12 hours of randomization HCQ was given. Standard dose of HCQ was 400 mg by mouth twice a day for day one followed by 200 mg 12 hourly for next 5 days.
Arm/Group | Standard of Care (SOC) | Intervention Group
Number analyzed (Participants) | 151 | 349
Participants | 5 | 11

2. Secondary Outcome: Viral Clearance
Description: PCR negativity on day 7 and 14 after admission
Time Frame: 14 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 days after first dose of HCQ or SOC
Description: Daily ECG, visual assessment, and Blood complete picture
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/349
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/349
Other Adverse Events (participants affected / at risk) | 0/151 | 0/349

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT04491994/Prot_SAP_000.pdf